CLINICAL TRIAL: NCT06326723
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Phase 1 Clinical Study to Investigate the Pharmacokinetics, Safety, and Tolerability After Single- and Multiple-Dose Daridorexant in Chinese Healthy Subjects
Brief Title: Investigate the PK, Safety, and Tolerability After Single and Multiple Dose Daridorexant in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0808-101
Record Dates: First submitted 2024-02-17; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25mg group (Experimental): Dose:25mg daridorexant or placebo Treatment Assignment :Day 1 SD, Day 4 - Day 8 MD (qdy) Number of subjects:16 (12 daridorexant + 4 placebo)
  Interventions: Drug: Daridorexant
- 50mg group (Experimental): Dose:50mg daridorexant or placebo Treatment Assignment :Day 1 SD, Day 4 - Day 8 MD (qdy) Number of subjects:16 (12 daridorexant + 4 placebo)
  Interventions: Drug: Daridorexant

INTERVENTIONS:
Drug: Daridorexant — 25 mg group: Daridorexant group: strength 25 mg, administered at a dose of 25 mg; administered orally under fasting conditions, single dosing on Day1, and daily dosing on Day 4-8.
  Placebo control group: administered in the same manner as the test drug.
  50 mg group: Daridorexant group: strength 50 mg, administered at a dose of 50 mg; administered orally under fasting conditions, single dosing on Day 1, and daily dosing on Day 4-8.
  Placebo control group: administered in the same manner as the test drug.
  Drug is to be administered at the same time every day, and the dosing window is recommended to be at 08:00 AM (±1 h) on the dosing day. Drinking water and other liquids should be avoided for 1 hour before and after dosing on the day of blood collection (except the water used to swallow the tablets.).

SUMMARY:
This clinical study is a single-center, randomized, double-blind, placebo-controlled Phase 1 clinical study to assess the PK characteristics and safety and tolerability of single and multiple dose daridorexant in 32 healthy adult Chinese subjects.

DETAILED DESCRIPTION:
This clinical study is a single-center, randomized, double-blind, placebo-controlled Phase 1 clinical study to assess the PK characteristics and safety and tolerability of single and multiple dose daridorexant in healthy adult Chinese subjects. This study will consist of a 20-day screening period, a 1-day baseline, a 11-day in patient period, and a 27-day follow-up period. The subjects will arrive at the study site on Day -1, and the subjects will be discharged from the study site on Day11.

32 healthy subjects (18-55 years) will be randomized. Two dose levels are planned (25 mg and 50 mg). 16 healthy subjects will be randomized with a ratio of 3:1 to receive 25mg daridorexant or matched placebo and another 16 healthy subjects will be randomized with a ratio of 3:1 to receive 50mg daridorexant or matched placebo. On Day 1, each subject will receive a single dose of daridorexant or placebo in the morning under fast conditions and PK samples will be collected up to 72 h post dose. Subject will receive repeated doses of daridorexant or placebo from day 4 to day 8 (QD) in the morning under fasting conditions and PK samples will be collected up to 72 h post last dose. The final follow-up visit will be conducted on Day 38, 30 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study. Signed informed consent in the local language prior to any study-mandated procedure.
2. Healthy Chinese male or female subjects aged between 18 and 55 years (inclusive) at screening.
3. Body Mass Index (BMI) ≥ 19 and ≤ 26 kg/m2, weight at least 45 kg for female, weight at least 50 kg for male at screening.
4. General good health at screening, with no abnormalities or abnormal clinically insignificant results based on medical history and physical examination, vital signs, laboratory tests, and 12-lead ECG performed at the time of screening. 50 bpm≤Resting heart rate (HR)≤100 bpm, 90mmHg <systolic blood pressure<140 mmHg or 50 mmHg<diastolic blood pressure<90 mmHg, ECG evidence of a QTcF interval of no more than 450 ms for male, ECG evidence of a QTcF interval of no more than 470 ms for female, (ECG monitors will be conducted for three times in five minutes, and mean values of three monitor results will be used)
5. Negative results from alcohol breath test and urine drug screen at Day -1.
6. Subjects (including male subjects) are willing to voluntarily use effective contraception from screening visit until 30 days after the end of the last dose and had no plans to become pregnant, planned parenthood or sperm/egg donation plans; Or subjects after surgical sterilization, or postmenopausal female subjects (female subjects with natural menopause ≥12 months can be considered postmenopausal; If age <50 years by follicle stimulating hormone level confirmed)

Exclusion Criteria:

1. Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
2. Intubation or repeat venipuncture is not appropriate.
3. Treatment with any prescription medications or over-the-counter medications (including herbal medicines) within 14 days prior to (first) study drug administration.
4. Have received any vaccine (including COVID-19 vaccine) prior to screening; have plan to receive vaccine (COVID-19 vaccine) during the study period or within 30 days after the last dose.
5. Not able or willing to stop treatment with moderate or strong cytochrome P450 (CYP)3A4 inhibitors, or treatment with moderate or strong CYP3A4 inducers, within 14 days prior to (first) study drug administration.
6. Not able or willing to stop consumption of grapefruit, Seville (bitter) oranges or juices from those fruits within 14 days prior to (first) study drug administration.
7. Treatment with another investigational drug within 3 months prior to screening or having participated in more than four investigational drug studies within 1 year prior to screening.
8. Use any nicotine or tobacco containing products (>5 cigarettes/day) within 3 years prior to day 1 and inability to refrain from smoking during the study.
9. Alcohol abuse（≥ 14 standard drinks units per week; 1 unit: 285 mL beer or 25 mL spirits or 100 mL wine） within 3 years prior to day 1 and inability to refrain from taking alcohol during the study.
10. Drinking excessive tea (>15 g tea leaves/day; 1 cup of tea contains about 3~5 g of tea leaves) or caffeine (>500 mg/ day, 1 cup of coffee contains about 85 mg of caffeine) and inability to refrain from drinking tea or caffeinated beverage during the study.
11. History or clinical evidence of any disease, and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of the study drugs (appendectomy and herniotomy allowed; cholecystectomy not allowed).
12. History of drug abuse.
13. Loss of 400 mL or more of blood, or an equivalent amount of plasma, within 3 months prior to screening.
14. Positive result to any of the following tests: HIV, hepatitis B, hepatitis C, and syphilis.
15. Known hypersensitivity to any excipients of the drug formulations.
16. Modified Swiss Narcolepsy Scale total score < 0 at screening. History of narcolepsy or cataplexy.
17. Any surgery planned during the study period.
18. Legal incapacity or limited legal capacity at screening
19. History of tuberculosis (TB).
20. Pregnant or lactating women, or positive pregnancy test results.
21. Any suicidal ideation with intent, with or without a plan (at screening):

    Planned or unplanned any suicidal thoughts; That is, answer yes to question 4 or 5 of the Suicidal ideation section of the lifetime version C-SSRS©. Lifetime past C-SSRS© Suicidal Behavior section indicates a history of suicide attempts.
22. Any circumstances or conditions which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Endpoints1 | Day1-Day11
  Maximum plasma concentration (Cmax)
Pharmacokinetic Endpoints2 | Day1-Day11
  Area under the concentration-time curve from zero to 24 hours (AUC0-24)
Pharmacokinetic Endpoints3 | Day1-Day11
  Aarea under the concentration-time curve from zero to 48 hours (AUC0-48)
Pharmacokinetic Endpoints4 | Day1-Day11
  Area under the concentration-time curve from zero to time t of the last measured concentration above the limit of quantification (AUC0-t)
Pharmacokinetic Endpoints5 | Day1-Day11
  area under the concentration-time curve from zero to infinity (AUC0-∞)
Pharmacokinetic Endpoints6 | Day1-Day11
  Time to reach maximum concentration (Tmax)
Pharmacokinetic Endpoints7 | Day1-Day11
  Terminal half-life (t1/2), and accumulation index (AI)

SECONDARY OUTCOMES:
Safety Endpoints1 | Day1-Day11
  Number and proportion of subjects with treatment-emergent adverse events
Safety Endpoints2 | Day1-Day11
  Number and proportion of subjects with treatment-emergent serious adverse events
Safety Endpoints3 | Day1-Day38
  Clinically significant vital sign abnormalities after the first dose of study drug up to 30 days after the last dose
Safety Endpoints4 | Day1-Day38
  Clinically significant physical examination abnormalities after the first dose of study drug up to 30 days after the last dose
Safety Endpoints5 | Day1-Day38
  Clinically significant blood routine test abnormalities after the first dose of study drug up to 30 days after the last dose
Safety Endpoints6 | Day1-Day38
  Clinically significant urinalysis abnormalities after the first dose of study drug up to 30 days after the last dose
Safety Endpoints7 | Day1-Day38
  Clinically significant abnormal blood biochemistry from the first dose of the study drug to 30 days after the last dose
Safety Endpoints8 | Day1-Day38
  Clinically significant ECG changes after the first dose of study drug up to 30 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No